CLINICAL TRIAL: NCT02483845
Title: Pilot Study of Natalizumab in the Treatment of Patients With Inclusion Body Myositis
Brief Title: Natalizumab in Inclusion Body Myositis (IBM)
Acronym: IBM-NAT
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Phoenix Neurological Associates, LTD (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBM-2013; 117571 (Other: IND approval)
Record Dates: First submitted 2013-05-31; First posted 2015-06-29 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Inclusion Body Myositis (IBM)
MeSH Terms: conditions — Myositis, Inclusion Body | interventions — Natalizumab

ARMS (1):
- Natalizumab (Experimental): Natalizumab therapy will be given at 300mg intravenously every 4 weeks for 24 weeks
  Interventions: Drug: Natalizumab

INTERVENTIONS:
Drug: Natalizumab
  Other Names: Tysabri

SUMMARY:
Muscle biopsies of patients with Inclusion Body Myositis (IBM) have demonstrated a T-cell predominant inflammatory infiltrate, therefore, new agents targeting T -cell mediated cell death may be a novel treatment for IBM. Such an agent capable of preventing T-cell movement out of the vasculature, such as natalizumab, may be beneficial in IBM patients. Six patients will be recruited to participate in this phase I trial.

DETAILED DESCRIPTION:
This is a phase I open label, non-placebo controlled trial evaluating the safety and efficacy of natalizumab in patients with IBM. Pre and post treatment muscle biopsies including measurements of the degree of inflammation as well as the types of inflammatory cells will be measured. The investigators will also assess quality of life, the inclusion body myositis functional rating score (IBM-FRS), and patient and physician global impression of change. Manual muscle testing and quantitative dynamometry will also be evaluated to see if patient's strength improves.

Patients who are eligible to participate and have signed a consent form will have a muscle biopsy performed at baseline and at the end of the study. Physical and neurological exams, as well as IBM-FRS, safety labs will be conducted and collected at monthly visits. Patients will start natalizumab therapy at 300mg intravenously every 4 weeks for 24 weeks. All study related procedures will be conducted at Phoenix Neurological Associates, as well as all infusions and muscle biopsies

ELIGIBILITY:
Inclusion Criteria:

1. Definite diagnosis of sporadic IBM through previous muscle biopsies
2. Age 21-85
3. FVC> 50%
4. Muscle function adequate for quantitative muscle testing
5. JC virus negative at screening

Exclusion Criteria:

1. Previous therapy with natalizumab.
2. Treatment with other immunosuppressive agents within the last 12 months
3. Quadriceps strength less than or equal to 2/5 at baseline
4. Known malignancy
5. Pregnancy or breastfeeding
6. History of abnormal laboratory results indicative of any significant medical disease that would preclude the use of natalizumab
7. Any clinically significant infectious illness in the 30 days before enrollment

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-05; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Determine if natalizumab is effective and safe in the treatment of patients with IBM (muscle biopsies) | 12 months
  muscle biopsies to determine inflammation
Determine if natalizumab is effective and safe in the treatment of patients with IBM (manual muscle testing) | 12 months
  MMT - manual muscle testing to determine strength

SECONDARY OUTCOMES:
Secondary outcome measures will involve an assessment of pre and post treatment muscle biopsies including measurements of the degree of inflammation as well as the types of inflammatory cells. (blood levels) | 12 months
  Safety labs - to determine blood levels
Secondary outcome measures will involve an assessment of pre and post treatment muscle biopsies including measurements of the degree of inflammation as well as the types of inflammatory cells. (pain scores) | 12 months
  Pain scores on a visual analog scale
Secondary outcome measures will involve an assessment of pre and post treatment muscle biopsies including measurements of the degree of inflammation as well as the types of inflammatory cells. (functional rating score scale) | 12 months
  IM-FRS a functional rating score scale

CONTACTS AND LOCATIONS:
Overall Officials: Todd Leveine, MD, Principal Investigator — Phoenix Neurological
Locations (1):
- Phoenix Neurological Insitutute, Phoenix, Arizona, United States